CLINICAL TRIAL: NCT01966016
Title: Efficacy and Safety of Multisite Cardiac Resynchronization Therapy - a Prospective Single Center Study in Selected Patient Population
Brief Title: Efficacy and Safety of Multisite Cardiac Resynchronization Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Arie Budovsky, CRA, Barzilai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRZ0046-12CTIL
Record Dates: First submitted 2013-08-26; First posted 2013-10-21 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Ventricular Tachycardia
Keywords: LV- Left Ventricular; CRT- Cardiac resynchronization therapy; MSCRT- Multisite Cardiac resynchronization therapy (P-pacemaker; D-defibrillator); BBB -bundle branch block
MeSH Terms: conditions — Tachycardia, Ventricular; Bundle-Branch Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- biventricular pacing (Experimental): The first configuration will be biventricular pacing (RV and postero-lateral branch of CS for LV pacing), as accepted
  Interventions: Procedure: Pacing
- triventricular pacing (Experimental): The second configuration will be triventricular pacing (RV+ postero-lateral branch of CS for LV pacing+ antero-lateral branch of CS for LV pacing) i.e. multisite LV pacing
  Interventions: Procedure: Pacing

INTERVENTIONS:
Procedure: Pacing — In this study we intend to include patients that have indication to and are intended to undergo CRT implantation with an additional electrode on LV, that have inclusion criteria and have signed an informed consent.
  In this study we will include 20 patients for each study arm (overall 100)- each patient will have both treatment configurations and these two will be compared

SUMMARY:
Cardiac resynchronization therapy (CRT) is a proven therapy in patients with severe left ventricular (LV) dysfunction with ejection fraction (EF)<35%., moderate to severe congestive heart failure and wide QRS in ECG. Positive response presents as improvement in quality of life, decrease in congestive hrat failure symptoms and signs, improvements in echocardiographic measurements and longer survival. About 30% of the patients do not respond to this treatment.

A decrease in clinical response to CRT is expected in patients with those predictors: advanced age, male, ischemic etiology of cardiomyopathy, Non-LBBB pattern in ECG, lack of mechanical dyssynchrony, large scar in LV, congestive heart failure stage IV, and non-cardiac co-morbidities (lung disease, pulmonary hypertension, renal failure and diabetes).

There are few solutions to increase the rate of clinical response to CRT, for example: endocardial pacing of LV or pacing a few simultaneous sites on LV. A study that investigated a method of simultaneous pacing on LV of patients with congestive heart failure and LBBB with QRS>150ms has shown major improvement of cardiac contraction (increased dP/dtmax) compared to a single pacing site over a postero-basal or lateral wall site).

Implantation of pacemaker leads- one in right ventricle (RV) and two over LV, i.e. multisite cardiac resynchronization therapy (MSCRT), has a few potential advantages, compared to conventional CRT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe LV dysfunction, severe heart failure (NYHA FC III-IV and at least one hospitalization for congestive heart failure in the past 3 months before inclusion) on optimal medical treatment and that have narrow complex QRS or RBBB. These patients have an indication for ICD implantation.
2. Patients with conventional indications for CRTD implantation and EF<25%, QRS>150ms and severe heart failure (NYHA FC>III).
3. Patients with an indication for pacemaker implantation and an expected high rate of pacing (complete AV block or prior to AVN ablation) and a wish to avoid RV pacing (example: severe TR).
4. Patients with refractory ventricular tachycardia and severe LV dysfunction (EF<35%) that continue to have VT episodes despite antiarrhythmic drugs and despite recurrent VT ablations. Those patients have indication for ICD.
5. Patients with conventional indications for CRT but during implantation the anatomy is such that the site of implantation is not optimal (QRS>200ms). In these cases we will add an electrode in the opposite branch of the coronary sinus.

Exclusion Criteria:

Pregnancy

* Patients included in another study
* Patients that have other solutions that could avoid implantation (medications, ablation, etc

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-11-20 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2015-11-17 (Actual)

PRIMARY OUTCOMES:
Multisite cardiac resynchronization therapy | 2 years
  In this research we intend to check the efficacy of MSCRT pacing mode in different populations of patients that are not yet included in the published guidelines.
  Primary end point: Immediate improvement in echo measurements of LVESV of the patient (Each patient is his own control. We expect 15% improvement versus baseline echo measurements or a difference of 5% from one measurements to another).

SECONDARY OUTCOMES:
decrease in arrhythmia burden | up to 1 year
  A clinical improvement regarding: decrease in arrhythmia burden, improvement in 6 minute walk results, decrease in number of hospitalizations, improvement in NYHA FC of at least one grade, and improvement in quality of life scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilai Medical Center, Ashkelon, Israel